CLINICAL TRIAL: NCT05904600
Title: Respiratory Muscle Training to Improve Functional Capacity and Prevent Respiratory Complications in Adults With Spinal Cord Injury
Brief Title: Respiratory Muscle Training in Adults With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FFEHNP
Record Dates: First submitted 2023-05-11; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Breathing exercises; Respiratory muscle training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Breathing Exercises; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masking of the researchers: randomisation of the sample will be performed using STATA software by a member of the research team who will not be involved in patient recruitment or data collection. The interventions will be carried out by researchers different from those who will perform the evaluation of the outcomes.
  Masking of the participants: the control group will have a training of the respiratory muscles simulated with the same device as the intervention group. They will use the device without load and with an opaque adhesive tape surrounding the device to mask the valve position.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training (Experimental): Respiratory muscle training with the Orygen-Dual Valve (Forumed S.L. ESP) and an initial load of 30% of their maximum inspiratory and expiratory pressures.
  Interventions: Device: Respiratory muscle training
- Control group (Sham Comparator): Simulated training with the Orygen-Dual Valve (Forumed S.L. ESP), without load.
  Interventions: Device: Control group

INTERVENTIONS:
Device: Respiratory muscle training — The training of the intervention group will have an initial workload of 30% of maximal inspiratory and expiratory pressures, which will be increased weekly by 10% according to tolerance, if not tolerated by 5%. In addition, patients will be instructed to maintain a normal respiratory rate (12-16 breaths per minute). Moreover, they will continue their usual treatment.
  Arms: Respiratory muscle training
Device: Control group — In the control group, the respiratory muscle training will be simulated by using the device without load throughout the study period using an opaque adhesive tape surrounding the device to mask the valve position.
  Arms: Control group

SUMMARY:
The purpose of this study is to investigate the effectiveness of a programme based on inspiratory and expiratory muscle training to improve respiratory muscle strength, functional capacity and avoid pulmonary complications in adults with cervical or high dorsal spinal cord injury (C5-D5) in acute phase.

DETAILED DESCRIPTION:
The design of the study is a randomised, triple-blind clinical trial with a control group.

The size of the sample will be 56 participants with cervical spinal cord injury and 56 with dorsal spinal cord injury. They will be randomized in two groups: experimental or control. The experimental group will perform combined inspiratory and expiratory muscle training as part of their rehabilitation programme during 6 weeks. The control group will continue their usual treatment.

Measurements will be taken at baseline, and post-intervention.

The statistical analysis will be an intention-to-treat analysis, and the data processing and analysis will be carried out with the Statistical Package for the Social Sciences (SPSS) version 24.0 for Windows (Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with spinal cord injury.
* Over 18 years of age.
* Time of evolution less than 6 months and at least 4 weeks after the date of injury.
* Level of lesion between C5 and D5 and degree of involvement A or B. In case of involvement A with partial preservation zone this should not include abdominal musculature according to the international standardised classification of the American Spinal Injury Association.

Exclusion Criteria:

* People with chest trauma.
* Mechanically ventilated.
* Pregnant women.
* Any medical or psychiatric condition that could affect the ability to complete the study.
* Carrying a tracheostomy tube that does not tolerate occlusion.
* People who can not sit upright.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in maximal expiratory pressure | Change after 6 weeks of intervention compared to baseline
  The measurement of maximum static respiratory pressures will consist of performing maximum forced inspiration and expiration manoeuvres against an occluded airway in order to measure the pressure generated in the mouth, using a manometer or a pressure transducer, since, with the glottis open, the pressure in the mouth must be equal to the alveolar pressure.
Change in maximal inspiratory pressure | Change after 6 weeks of intervention compared to baseline
  The measurement of maximum static respiratory pressures will consist of performing maximum forced inspiration and expiration manoeuvres against an occluded airway in order to measure the pressure generated in the mouth, using a manometer or a pressure transducer, since, with the glottis open, the pressure in the mouth must be equal to the alveolar pressure.

SECONDARY OUTCOMES:
Change in forced vital capacity (FVC) | Change after 6 weeks of intervention compared to baseline
  Using a spirometer, with the mouthpiece tightly sealed around the lips, the participant is asked, from the residual volume, to perform a rapid but unforced maximal inspiratory manoeuvre. With an apnoea of less than one second at total lung capacity, the participant is asked to exhale maximally, rapidly and forcibly, until the lungs are completely empty. At this point, the participant is strongly encouraged to start the manoeuvre abruptly and to prolong the exhalation long enough to reach RV.
Change in coughing capacity | Change after 6 weeks of intervention compared to baseline
  Measurement of cough capacity will be performed by determining peak cough flow using a peak expiratory flow meter (Mini Wright flow meter; Clement Clarke International Ltd., Essex, UK).
Change in elbow flexion strength | Change after 6 weeks of intervention compared to baseline
  In all subjects, the maximum load they can move in one repetition (1RM) in both limbs will be assessed for elbow flexion with Microfet4 dynamometer; Hoggan Health Industries, West Jordan, Utah.
Change in shoulder flexion strength | Change after 6 weeks of intervention compared to baseline
  In all subjects, the maximum load they can move in one repetition (1RM) in both limbs will be assessed for shoulder flexion with Microfet4 dynamometer; Hoggan Health Industries, West Jordan, Utah.
Change in number of people with respiratory complications | Change after 6 weeks of intervention compared to baseline
  Respiratory complications will be assessed by consulting the medical history.
Change in health-related quality of life assessed by Short-Form 36 questionnaire. | Change after 6 weeks of intervention compared to baseline
  Health-related quality of life will be measured with the Short-Form 36 questionnaire, with values ranging from 0 to 100 (higher scores mean better health-related quality of life).
Change in forced expiratory volume in the first second (FEV1) | Change after 6 weeks of intervention compared to baseline
  Using a spirometer, with the mouthpiece tightly sealed around the lips, the participant is asked, from the residual volume, to perform a rapid but unforced maximal inspiratory manoeuvre. With an apnoea of less than one second at total lung capacity, the participant is asked to exhale maximally, rapidly and forcibly, until the lungs are completely empty. At this point, the participant is strongly encouraged to start the manoeuvre abruptly and to prolong the exhalation long enough to reach RV.
Change in cardiorespiratory fitness | Change after 6 weeks of intervention compared to baseline
  Cardiorespiratory fitness will be measured using the 6-minute wheelchair propulsion test (adapted from Bass A et al. 2020). This is a validated test to measure cardiorespiratory fitness through a submaximal exercise test where the patient performs a 25-metre figure-eight run for 6 minutes and the distance covered in that time is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Torres-Costoso, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Sara Reina Gutiérrez, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
Only the research team, and the health authorities, who have a duty of confidentiality, will have access to all data collected by the study. Information that cannot be identified may be passed on to third parties.